CLINICAL TRIAL: NCT06119633
Title: Immediate Tissue Expander and Lipofilling After Mastectomy for Breast Cancer Recurrence Following Lumpectomy and Irradiation: Retrospective Multicentric Clinical Trial
Brief Title: Implant-based Breast Reconstruction and Mastectomy With Fat Grafting After Breast Conserving Surgery and Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Morgagni Pierantoni Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 217/23
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Radiotherapy; Implant-based breast reconstruction; Fat grafting; Adipose tissue transplant; Lipofilling; Hodgkin lymphoma; Expander
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immediate tissue expander and fat grafting after mastectomy (Experimental): Patients underwent simple mastectomy, skin-sparing or nipple-sparing mastectomy and implant-based, two-stage breast reconstruction: contextual mastectomy and expander positioning were performed during first stage (stage I) while substitution of the expander with definitive implant occurred during second stage (stage II). Fat grafting with regenerative intent was performed during stage I or between stage I and II. Adipose tissue was harvested from the abdomen, flanks, trochanter regions, inner thigh and medial aspect of knees. Fat was injected in the subfascial plane of the pectoralis major muscle with blunt cannula in order to avoid thrombo-embolic risks. At least six months after stage I patients underwent expander substitution with definitive implant and contralateral mammoplasty when required. In case of complications that required removal of the implant, autologous reconstruction was performed.
  Interventions: Procedure: Immediate tissue expander and lipofilling after mastectomy

INTERVENTIONS:
Procedure: Immediate tissue expander and lipofilling after mastectomy — Implant-based breast reconstruction and fat grafting after salvage or prophylactic mastectomy in patients previously exposed to radiation therapy on the breast as adjuvant treatment after breast conserving surgery (BCS) or on thoracic wall for Hodgkin Lymphoma (HL).

SUMMARY:
Higher rates of complications and poorer cosmetic outcomes have been reported after salvage mastectomy and implant-based versus autologous reconstruction in patients previously exposed to radiation therapy (i) on the breast as adjuvant treatment after breast conserving surgery (BCS) or (ii) on thoracic wall for Hodgkin Lymphoma (HL). Nevertheless, selected patients with favourable preoperative soft-tissue assessment may benefit from alloplastic reconstruction and fat grafting that has been suggested as an effective technique to promote the regeneration of irradiated tissues.

The aims of this study are to assess:

1. the feasibility of implant-based breast reconstruction and fat grafting after mastectomy (simple mastectomy, nipple-sparing and skin-sparing mastectomy)
2. oncological safety of implant-based breast reconstruction and fat grafting.

DETAILED DESCRIPTION:
National Comprehensive Cancer Network guidelines recommend autologous reconstruction as the preferred breast reconstruction after mastectomy in previously irradiated patients because of higher complication rates and worse aesthetic outcomes as compared to immediate breast implant reconstruction. In fact, unacceptable rates of complications (60-70%) have been reported by first experiences. Instead, autologous reconstruction showed lower complication rates as compared to implant-based breast reconstruction (25.5% vs 50.9%). However, it may not be indicated in patients with previous surgery at the donor site or in case of other contraindications, requires longer surgical time and is at risk of donor-site morbidity and loss of sensation.

On the other hand, fat grafting improves softness of tissues and scars, releasing their rigidity and for these effects it has been studied for effectively promoting the regeneration of irradiated tissues, enlarging the envelope thickness for safety reasons, optimizing cosmetic outcomes and ultimately increasing patient comfort and quality of life.

Therefore, a surgical technique combining implant-based breast reconstruction after mastectomy and fat grafting may favor alloplastic reconstruction in selected patients.

The investigators enroll patients candidate to mastectomy and breast reconstruction who had received prior adjuvant radiation therapy after breast conserving surgery (BCS) or radiation therapy for the treatment of Hodgkin Lymphoma (HL).

Aims of the study are to investigate (i) the feasibility of implant-based breast reconstruction and fat grafting after mastectomy (simple mastectomy, nipple-sparing and skin-sparing mastectomy); (ii) the oncological safety of implant-based breast reconstruction and fat grafting.

ELIGIBILITY:
Inclusion Criteria:

* patients candidate to mastectomy (salvage mastectomy for breast cancer recurrence or prophylactic mastectomy) who had been irradiated as adjuvant treatment after breast conserving surgery or as treatment for Hodgkin lymphoma
* signed informed consent to participate and to implant-based breast reconstruction
* absence of distant metastases or other malignancies.

Exclusion Criteria:

- presence of distant metastases or other malignancies.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Complication rates after stage I and II | 1 month, 6 months and 12 months
  Identification of complication rates after stage I and II, measuring percentage of complications (pain and patient discomfort, partial necrosis of mastectomy flaps, nipple-areolar necrosis, delayed wound healing, capsular contracture, bleeding, expander or implant exposition, infection, expander rupture, re-operations, reconstruction failures) over the total number of surgical procedures of stage I and II.
Patient's satisfaction | 12 months
  Self-assessed patient reports for identification of patient's satisfaction, measuring percentage of patients that were satisfied with results overall.
Cosmetic outcomes | 1 month, 6 months and 12 months
  Clinical and photography-based assessments for cosmetic outcomes measurement graded by a plastic breast surgeon as excellent, very good, good, fair, or poor.

SECONDARY OUTCOMES:
Oncological safety of implant-based breast reconstruction and fat grafting. | 5 years
  Identification of rate of loco-regional and distant metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Listorti, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy; Secondo Folli, MD, Study Director — Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
Locations (2):
- Italy (2):
  - Morgagni Pierantoni Hospital, Forlì
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan

REFERENCES:
- [Result] Krueger EA, Wilkins EG, Strawderman M, Cederna P, Goldfarb S, Vicini FA, Pierce LJ. Complications and patient satisfaction following expander/implant breast reconstruction with and without radiotherapy. Int J Radiat Oncol Biol Phys. 2001 Mar 1;49(3):713-21. doi: 10.1016/s0360-3016(00)01402-4. PMID 11172953
- [Result] Dickson MG, Sharpe DT, Dickson WA, Wilde GP, Brennan TG, Roberts AH. Breast reconstruction by tissue expansion. Ann R Coll Surg Engl. 1987 Jan;69(1):19-21. PMID 3566111
- [Result] Manyam BV, Shah C, Woody NM, Reddy CA, Weller MA, Juloori A, Naik M, Valente S, Grobmyer S, Durand P, Djohan R, Tendulkar RD. Long-Term Outcomes After Autologous or Tissue Expander/Implant-Based Breast Reconstruction and Postmastectomy Radiation for Breast Cancer. Pract Radiat Oncol. 2019 Nov;9(6):e497-e505. doi: 10.1016/j.prro.2019.06.008. Epub 2019 Jun 22. PMID 31238166
- [Result] Khansa I, Boehmler JH 4th. Aesthetic outcomes in women undergoing breast-conserving therapy followed by mastectomy and microsurgical reconstruction. Microsurgery. 2015 Jan;35(1):21-8. doi: 10.1002/micr.22225. Epub 2014 Jan 21. PMID 24449018
- [Result] Debald M, Pech T, Kaiser C, Keyver-Paik MD, Walgenbach-Bruenagel G, Kalff JC, Kuhn W, Walgenbach KJ. Lipofilling effects after breast cancer surgery in post-radiation patients: an analysis of results and algorithm proposal. Eur J Plast Surg. 2017;40(5):447-454. doi: 10.1007/s00238-017-1311-1. Epub 2017 May 29. PMID 28989237
- [Result] Salgarello M, Visconti G, Barone-Adesi L. Fat grafting and breast reconstruction with implant: another option for irradiated breast cancer patients. Plast Reconstr Surg. 2012 Feb;129(2):317-329. doi: 10.1097/PRS.0b013e31822b6619. PMID 21987041
- [Result] Coleman SR, Saboeiro AP. Fat grafting to the breast revisited: safety and efficacy. Plast Reconstr Surg. 2007 Mar;119(3):775-85; discussion 786-7. doi: 10.1097/01.prs.0000252001.59162.c9. PMID 17312477
- See also: last day of access July 26th 2023 — https://www.nccn.org/professionals/physician_gls/pdf/breast.pdf